CLINICAL TRIAL: NCT06051058
Title: Care Transitions App for Patients With Multiple Chronic Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lipika Samal, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P001447
Record Dates: First submitted 2023-09-18; First posted 2023-09-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Congestive Heart Failure; Diabetes; Diabetes Mellitus; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The design is a randomized trial with patients recruited inpatient from Brigham and Women's Hospital and nested within primary care practices in the MGB healthcare system. The unit of randomization is the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Care Transitions App (Experimental): Use of the Care Transitions App to support the care transition for patients hospitalized and discharged with multiple chronic conditions will be compared to usual care.
  Interventions: Behavioral: Care Transitions App
- No Intervention: Usual Care (No Intervention): Usual care transition care for patients hospitalized and discharged with multiple chronic conditions.

INTERVENTIONS:
Behavioral: Care Transitions App — Patients in the intervention arm will be randomized to receive the Care Transitions App and utilize it to support their care transition care plan for multiple chronic conditions.
  Arms: Experimental: Care Transitions App

SUMMARY:
The objective of this study is to widely implement and evaluate the Care Transitions App in a randomized controlled trial. The app the investigators designed for patients with multiple chronic conditions has four envisioned modules: 1) falls-reduction content, 2) a digital post-discharge transitional care plan (e.g., after hospital care plan, including education, medications, follow-up appointments, warning signs to watch for, nutrition, and other care plan activities), 3) a new module for patients with MCC (diabetes, congestive heart failure, and chronic kidney disease) including condition-specific post-discharge care plans with relevant symptom management activities, 4) a new post-discharge report module which summarizes key care transition findings and allows for patients to enter notes and questions for their providers and their own goals for recovery.

DETAILED DESCRIPTION:
Care transitions are a vulnerable period for patients, leading to a 20% rate of readmissions, 11% rate of post-discharge adverse drug events, 15% rate of falls, and 29% rate of total post-discharge adverse events. Hospital discharge for patients with multiple chronic conditions (MCC) is a challenge for the hospital care teams, primary care providers (PCPs) and patients/caregivers who face the challenge of complex medication regimens, as well as patient-specific challenges in fall prevention strategies. Specific challenges include poor communication among inpatient providers, patients, and ambulatory providers, poor quality and timeliness of discharge documentation, suboptimal patient understanding of post-discharge plans of care and their ability to carry out these plans, medication discrepancies and non-adherence after discharge, failure to follow up the results of tests pending at time of discharge, failure to schedule necessary ambulatory appointments, tests, and procedures, and lack of timely follow-up with ambulatory providers.

These risks are especially important for people living with multiple chronic conditions (PLWMCC), such as diabetes (DM), congestive heart failure (CHF), and chronic kidney disease (CKD). Each of these conditions requires a complex medication regimen which is often altered during the hospital admission. Often, the medications cannot be changed back to their original dose at the time of discharge because patients are eating less than usual, have become dehydrated, and their kidney function has been affected by nephrotoxic medications. Clearance of medications such as insulin is also altered and limited physical activity in the hospital places patients at increased risk for falls after discharge. All of these factors increase the risk of adverse events in the post-discharge period. An overarching goal of the intervention is to overcome common care transition challenges by simplifying the information patients and caregivers receive and empowering them to carry out their care plans.

Previous research supports the use of mobile apps for improving health outcomes among those living with chronic illness. While many apps are available for chronic disease management, most of them focus on a single chronic illness such as diabetes or heart failure, or self-management area such as medication management, sleep, or pain and do not specifically target the period of transition from hospital to home. The intervention will fill an existing gap by developing, rigorously testing, and disseminating a comprehensive Care Transitions App for patients with MCC that will provide comprehensive care transition information for disease self-management, medication safety, and fall prevention in a format that is simple and actionable.

The investigators will conduct a pragmatic randomized controlled trial in an academic medical center (Brigham and Women's Hospital) and primary care clinics to test the effectiveness of the Care Transitions App enrolling patients age 55 or older with MCC including Diabetes, congestive heart failure, and/or chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (55+) with a Brigham PCP or appointment in one of the 15 locations discharging from a BWH general medicine unit
* Discharging to home, home health care service or assisted living
* Fluent in spoken English in patient or healthcare proxy
* Patients with at least one of the conditions listed below + one additional chronic condition on the problem list.
* Patient with heart failure on the problem list
* Patient with type 2 diabetes on the problem list
* Patient with chronic kidney disease on the problem list

Exclusion Criteria:

* Adult patients (55+) with Westwood, Pembroke, or Transition Clinic PCP admitted to ICU, OBGYN, Surgical, Cardiology, Oncology, Orthopedics, or other Specialty Unit
* Pregnant
* Prisoner, institutionalized individual or in police custody
* Discharge planned within 3 hours of screening
* Patient too ill to participate or with active psychosis/serious mental illness, delirium, or severe dementia
* Not fluent in spoken English in patient and health proxy
* Unlikely to be discharged to home
* Lacks a device capable of accessing the app
* Lack of a working telephone for 30-day follow-up

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 798 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of the Care Transitions App on post-discharge adverse events | 30 Days
  Overall rate of post-discharge adverse events

SECONDARY OUTCOMES:
To determine the effect of the Care Transitions App on the 30-day readmission rate | 30 Days
  30-day readmission rate

CONTACTS AND LOCATIONS:
Overall Officials: Lipika Samal, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.